CLINICAL TRIAL: NCT01096927
Title: Non Operative Treatment for Acute Appendicitis: Study on Efficacy and Safety of Antibiotic Treatment (Amoxicillin and Clavulanic Acid) in Patients With Right Sided Lower Abdominal Pain
Brief Title: Non Operative Treatment for Acute Appendicitis
Acronym: NOTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maggiore Bellaria Hospital, Bologna (Other)
Responsible Party: Gregorio Tugnoli, Emergency and Trauma Surgery Unit, Department of Emergency, Maggiore Hospital Trauma Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 09079
Record Dates: First submitted 2010-03-29; First posted 2010-03-31 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-01

CONDITIONS: Lower Abdominal Pain; Right Iliac Fossa Pain; Acute Appendicitis
Keywords: Lower Abdominal Pain; Right Iliac Fossa Pain; Acute Appendicitis; Antibiotic Therapy; Conservative Management; Appendectomy; Recurrence; Length of hospital stay; Sick leave time; Short and Long Term Abdominal pain evaluation
MeSH Terms: conditions — Appendicitis; Recurrence | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non operative Treatment group (Experimental): Patients with Lower Abdominal and suspected Acute Appendicitis, treated non-operatively with 7 days antibiotic therapy (Amoxicillin and Clavulanic Acid)
  Interventions: Drug: Amoxicillin and Clavulanic Acid

INTERVENTIONS:
Drug: Amoxicillin and Clavulanic Acid — 7 days antibiotic therapy with Amoxicillin and Clavulanic Acid, 1 gr 3 times daily PO

SUMMARY:
Case control studies that randomly assign patients to either surgical or non-surgical treatment yield a relapse rate of approximately 14% at one year. It would be useful to know the relapse rate of patients who have, instead, been selected for a given treatment based on a thorough clinical evaluation, including physical examination and laboratory results (all characteristics forming the Alvarado Score) as well as radiological exams if needed or deemed helpful. If this clinical evaluation is useful,the investigators would expect patient selection to be better than chance, and relapse rate lower than 14%. Once the investigators have established the utility of this evaluation, the investigators can begin to identify those components that have predictive value (such as blood chemistry analysis, or CT findings). This is the first step toward developing an accurate diagnostic-therapeutic algorithm which will avoid the risks and costs of needless surgery.

This will be a single-cohort prospective interventional study. It will not interfere with the usual procedures, consisting of clinical examination in the Emergency Department (ED) and execution of the following exams at the physician's discretion: complete blood count with differential, C reactive protein, abdominal ultrasound, abdominal CT. Patients admitted to Emergency Department with Lower Abdominal and suspicion of Acute Appendicitis not needing immediate surgery, are requested by informed consent to undergo observation and non operative treatment with antibiotic therapy (Amoxicillin and Clavulanic Acid). The patients by protocol should not have received any previous antibiotic treatment during the same clinical episode. Patients not undergoing surgery will be physically examined 5 days later. During this follow-up visit, the patient will be given information about the study, will be invited to participate, and will be asked to sign an informed consent form. If the patient is under the age of 18 years, consent will be obtained from a parent or other legal guardian.

Telephone (or email) follow-ups will be conducted at 15 days, 6 months, and 12 months (see attached schedule) to monitor the state of the illness.

DETAILED DESCRIPTION:
Background: Acute appendicitis is one of the most common urgent conditions seen in general surgery practice. Complications can be severe and include perforation and generalized peritonitis. Traditionally, surgical appendectomy has been the primary treatment, even in cases of unconfirmed diagnosis, given the low incidence of major complications. In 15-30% of cases, in fact, the appendix is found to be free of disease upon resection. This procedure, however, is not without risk. It is associated with surgical wound infection, intestinal obstruction due to adhesions, pneumonia, and tubal infertility in females. For this reason, the possibility of using conservative treatment merits investigation. There is considerable debate regarding the utility of conservative treatment over surgical treatment in some cases of acute appendicitis, as few studies have addressed this issue to date. If deemed useful, it will become of utmost importance to make an accurate diagnosis and assessment in every patient in order to select the most appropriate treatment.

Hansson et al conducted a randomized clinical trial investigating the efficacy of conservative treatment compared to surgery for acute appendicitis. They reported that conservative treatment with antibiotics was efficacious in 91% of cases, with a 14% relapse rate at 12 month follow-up. One third of relapses occurred within the first 10 days of hospital discharge, while most of the remaining two thirds occurred between 3 and 16 months following discharge. The rates of minor complications such as diarrhea, vomiting, and nosocomial infections were similar among patients treated conservatively and those treated surgically. The incidence of major complications such as appendiceal abscess, paralytic ileus and pulmonary embolism, however, was significantly higher in those treated surgically (p<0.05).

A recent prospective randomized study conducted by Ajaz and colleagues compared antibiotic therapy to appendectomy in acute appendicitis. The authors reported that conservative treatment was not only safe and efficacious, but caused the patients less pain than did surgery, reducing the need for analgesic therapy (p<0.001). Ten percent of conservatively treated patients relapsed within 12 months of discharge.

A multicenter randomized trial conducted in Sweden yielded similar results: the rate of relapse in antibiotic treated patients was 14% at one year after discharge. Interestingly, this was equal to the rate of post-operative complications in patients treated surgically.

Based on these reports, conservative treatment seems to represent a valid therapeutic approach to acute appendicitis. Relapse rate is low and comparable to the rate of surgical complications.

Rationale: Case control studies that randomly assign patients to either surgical or non-surgical treatment yield a relapse rate of approximately 14% at one year. It would be useful to know the relapse rate of patients who have, instead, been selected for a given treatment based on a thorough clinical evaluation, including physical examination and laboratory results (all characteristics forming the Alvarado Score) as well as radiological exams if needed or deemed helpful. If this clinical evaluation is useful, the investigators would expect patient selection to be better than chance, and relapse rate lower than 14%. Once the investigators have established the utility of this evaluation, the investigators can begin to identify those components that have predictive value (such as blood chemistry analysis, or CT findings). This is the first step toward developing an accurate diagnostic-therapeutic algorithm which will avoid the risks and costs of needless surgery.

Study Description: This will be a single-cohort prospective interventional study. It will not interfere with the usual procedures, consisting of clinical examination in the Emergency Department (ED) and execution of the following exams at the physician's discretion: complete blood count with differential, C reactive protein, abdominal ultrasound, abdominal CT. Patients admitted to Emergency Department with Lower Abdominal and suspicion of Acute Appendicitis not needing immediate surgery, are requested by informed consent to undergo observation and non operative treatment with antibiotic therapy (Amoxicillin and Clavulanic Acid). The patients by protocol should not have received any previous antibiotic treatment during the same clinical episode. Patients not undergoing surgery will be physically examined 5 days later. During this follow-up visit, the patient will be given information about the study, will be invited to participate, and will be asked to sign an informed consent form. If the patient is under the age of 18 years, consent will be obtained from a parent or other legal guardian.

Telephone (or email) follow-ups will be conducted at 15 days, 6 months, and 12 months (see attached schedule) to monitor the state of the illness. The patient will be asked if he/she has undergone surgery since the first visit (5 days post-ED). If not, the patient will be asked:

1. has your illness improved, stayed the same, or worsened since its onset?
2. have you done any further tests or had additional doctor's visits for your illness?
3. after your initial emergency department visit, how much time did it take to return to your normal activities (physical activity, work, etc)? In the case of patients under the age of 18 years, the phone interview will be conducted with a parent or legal guardian.

Study Objectives:

Main Objective: Evaluate the outcome of patients treated conservatively, assessing the reliability of the initial clinical evaluation in predicting which conservatively-treated patients should have treated surgically.

Primary Outcomes are the following:

1. Short Term Efficacy of Antibiotic Treatment: Failure of the conservative treatment with antibiotic within the period of the Amoxicillin + Clavulanic Acid therapy (7 days), defined as readmission for abscence of clinical improvement and/or worsening abdominal pain and/or localized/diffuse peritonitis
2. Long Term Efficacy of Antibiotic Treatment: Efficacy of antibiotic therapy for acute appendicitis defined as incidence of recurrences of clinical episodes of appendicitis up to 1 year follow up
3. Long Term Efficacy of Antibiotic Treatment (NO need for surgery): Efficacy of antibiotic therapy for acute appendicitis defined as definite improvement without need for surgery within 1 year follow up
4. Safety of Antibiotic treatment: Major side effects/complications drug/treatment-related (i.e. Allergy or other complications treatment related such as abscess formation)

Secondary Outcomes are:

1. Minor Complications: Minor side effects/complications drug/treatment-related (i.e. bloating, diarrhea, gas, headache, heartburn, nausea, and vomiting)
2. Abdominal Pain after discharge: Assessment of abdominal pain / discomfort evaluated by mean of Numerical rating scale (NRS)
3. Length of Hospital stay: Length of clinical observation as inpatient
4. Outpatient clinic checkup: Number of follow up appointments scheduled in outpatient clinic
5. Sick Leave: Number of days of sick leave needed by the patient
6. Cost analysis: Analysis of the costs, including Antibiotic course, Length of Hospital Stay, Outpatient Clinic follow up appointments, sick leave days

Additional Objective: Identify clinical, laboratory or imaging findings that are predictive of relapse and need for appendectomy.

Study Design: Single cohort prospective interventional study. No experimental interventions or treatments will be employed beyond routine clinical care.

Inclusion Criteria: Any patient, male or female, above the age of 14 years (non-pediatric), who returns for the follow-up visit 5 days after the ED visit and consents participation between January 1, 2010 and December 31, 2010.

The investigators estimate a sample size of 160, the number of patients with suspected acute appendicitis we typically receive yearly in the ED.

Means of follow-up assessment: telephone interview (or e-mail)

ELIGIBILITY:
Inclusion Criteria:

1. Age >14 years
2. Lower / RIF Abdominal Pain
3. Clinical Suspicion of Acute Appendicitis:

   i.e.
   * Alvarado Score 5-6 (equivocal for acute appendicitis)
   * Alvarado Score 7-8 (probably appendicitis)
   * Alvarado Score 9-10 (highly likely appendicitis)
4. Informed consent (patient or legal representative)

Exclusion Criteria:

1. Diffuse peritonitis
2. Antibiotic (Penicillin) documented allergy
3. Ongoing previously started antibiotic therapy
4. Previous appendectomy
5. Positive pregnancy test
6. IBD history or suspicion of IBD recrudescence

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Short Term Efficacy of Antibiotic Treatment | within 7 days (Antibiotic treatment course)
  Failure of the conservative treatment with antibiotic within the period of the Amoxicillin + Clavulanic Acid therapy (7 days), defined as readmission for abscence of clinical improvement and/or worsening abdominal pain and/or localized/diffuse peritonitis
Long Term Efficacy of Antibiotic Treatment | 1 year
  Efficacy of antibiotic therapy for acute appendicitis defined as incidence of recurrences of clinical episodes of appendicitis up to 1 year follow up (at 15 days, 6 months, 1 year)
Long Term Efficacy of Antibiotic Treatment (NO need for surgery) | 1 year
  Efficacy of antibiotic therapy for acute appendicitis defined as definite improvement without need for surgery within 1 year follow up (at 15 days, 6 months, 1 year)
Safety of Antibiotic treatment | 7 days
  Major side effects/complications drug/treatment-related (i.e. Allergy or other complications treatment related such as abscess formation)

SECONDARY OUTCOMES:
Minor Complications | 15 days
  Minor side effects/complications drug/treatment-related (i.e. bloating, diarrhea, gas, headache, heartburn, nausea, and vomiting) (at 7 days, 15 days)
Abdominal Pain after discharge | 15 days
  Assessment of abdminal pain / discomfort evaluated by mean of Numerical rating scale (NRS) (at 7 days, 15 days)
Length of Hospital stay | 7 days
  Length of clinical observation as inpatient
Outpatient clinic checkup | 15 days
  Number of follow up appointments scheduled in outpatient clinic
Sick Leave | 1 year
  Number of days of sick leave needed by the patient (assessed at 7 days, 15 days, 6 months, 1 year)
Cost analysis | 1 year
  Analysis of the costs, including Antibiotic course, Length of Hospital Stay, Outpatient Clinic follow up appointments, sick leave days

CONTACTS AND LOCATIONS:
Overall Officials: Gregorio Tugnoli, MD, Study Chair — Emergency and Trauma Surgery Unit, Department of Emergency, Maggiore Hospital; Gregorio Tugnoli, MD, Study Director — Emergency and Trauma Surgery Unit, Department of Emergency, Maggiore Hospital; Nicola Antonacci, MD, Study Director — Emergency and Trauma Surgery Unit, Department of Emergency, Maggiore Hospital; Salomone Di Saverio, MD, Study Director — Emergency and Trauma Surgery Unit, Department of Emergency, Maggiore Hospital; Franco Baldoni, MD, Study Director — Emergency and Trauma Surgery Unit, Department of Emergency, Maggiore Hospital; Andrea Biscardi, MD, Principal Investigator — Emergency and Trauma Surgery Unit, Department of Emergency, Maggiore Hospital; Silvia Villani, MD, Principal Investigator — Emergency and Trauma Surgery Unit, Department of Emergency, Maggiore Hospital; Eleonora Giorgini, MD, Principal Investigator — Emergency and Trauma Surgery Unit, Department of Emergency, Maggiore Hospital; Gianluca Senatore, MD, Principal Investigator — Emergency and Trauma Surgery Unit, Department of Emergency, Maggiore Hospital; Nicola Clemente, MD, Principal Investigator — Emergency and Trauma Surgery Unit, Department of Emergency, Maggiore Hospital
Locations (1):
- Maggiore Bellaria Hospital, Bologna, Italy

REFERENCES:
- [Background] Malik AA, Bari SU. Conservative management of acute appendicitis. J Gastrointest Surg. 2009 May;13(5):966-70. doi: 10.1007/s11605-009-0835-5. Epub 2009 Mar 10. PMID 19277796 (Retraction: PMID 21975685 J Gastrointest Surg. 2011 Dec;15(12):2302)
- [Background] Deutsch AA, Shani N, Reiss R. Are some some appendectomies unnecessary? An analysis of 319 white appendices. J R Coll Surg Edinb. 1983 Jan;28(1):35-40. No abstract available. PMID 6834311
- [Background] Pieper R, Kager L, Nasman P. Acute appendicitis: a clinical study of 1018 cases of emergency appendectomy. Acta Chir Scand. 1982;148(1):51-62. No abstract available. PMID 7136412
- [Background] Styrud J, Eriksson S, Nilsson I, Ahlberg G, Haapaniemi S, Neovius G, Rex L, Badume I, Granstrom L. Appendectomy versus antibiotic treatment in acute appendicitis. a prospective multicenter randomized controlled trial. World J Surg. 2006 Jun;30(6):1033-7. doi: 10.1007/s00268-005-0304-6. PMID 16736333
- [Background] Eriksson S, Granstrom L. Randomized controlled trial of appendicectomy versus antibiotic therapy for acute appendicitis. Br J Surg. 1995 Feb;82(2):166-9. doi: 10.1002/bjs.1800820207. PMID 7749676
- [Background] Hansson J, Korner U, Khorram-Manesh A, Solberg A, Lundholm K. Randomized clinical trial of antibiotic therapy versus appendicectomy as primary treatment of acute appendicitis in unselected patients. Br J Surg. 2009 May;96(5):473-81. doi: 10.1002/bjs.6482. PMID 19358184
- [Derived] Di Saverio S, Sibilio A, Giorgini E, Biscardi A, Villani S, Coccolini F, Smerieri N, Pisano M, Ansaloni L, Sartelli M, Catena F, Tugnoli G. The NOTA Study (Non Operative Treatment for Acute Appendicitis): prospective study on the efficacy and safety of antibiotics (amoxicillin and clavulanic acid) for treating patients with right lower quadrant abdominal pain and long-term follow-up of conservatively treated suspected appendicitis. Ann Surg. 2014 Jul;260(1):109-17. doi: 10.1097/SLA.0000000000000560. PMID 24646528
- [Derived] Tugnoli G, Giorgini E, Biscardi A, Villani S, Clemente N, Senatore G, Filicori F, Antonacci N, Baldoni F, De Werra C, Di Saverio S. The NOTA study: non-operative treatment for acute appendicitis: prospective study on the efficacy and safety of antibiotic treatment (amoxicillin and clavulanic acid) in patients with right sided lower abdominal pain. BMJ Open. 2011 Feb 23;1(1):e000006. doi: 10.1136/bmjopen-2010-000006. PMID 22021722